CLINICAL TRIAL: NCT05545098
Title: The Role of Musculoskeletal Ultrasound Versus Serum Survivin and Lubricin Levels in Evaluation of Disease Activity in Juvenile Idiopathic Arthritis
Brief Title: MSUS Versus Serum Survivin and Lubricin Levels in Evaluation of Disease Activity in JIA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yostina Ramzy Gadallah Ghattas, doctor, Assiut University
Other Study IDs: Juvenile idiopathic arthritis
Record Dates: First submitted 2022-09-03; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JIA patients: * Assessment of Survivin and Lubricin in the serum and in the Synovial fluid if available in JIA patients
  * Assessment of activity using Juvenile arthritis disease activity score in 27 joints (JADAS 27) in the studied JIA patients.
  * Identifying the prevalence of functional disability in JIA children and adolescents using the childhood health assessment questionnaire (CHAQ).
  * performing MSUS on the involved joints.
- control group: Assessment of Survivin and Lubricin in the serum

SUMMARY:
Aim of the work The aim of this study is to compare the role of musculoskeletal ultrasound to serum Survivin and Lubricin in detection of disease activity in patients with oligoarticular and polyarticular juvenile idiopathic arthritis.

Objectives

* To assess disease activity using Juvenile arthritis disease activity score in 27 joints (JADAS 27) in the studied JIA patients.
* To identify the prevalence of functional disability in JIA children and adolescents using the childhood health assessment questionnaire (CHAQ).
* To perform MSUS on the involved joints.
* To assess Survivin in the serum and in the synovial fluid if available in JIA patients.
* To assess Lubricin in the serum and in the synovial fluid if available in JIA patients.
* To compare the disease activity across individual patients using JADAS 27, MSUS and their relation to serum level of Survivin and lubricin.

DETAILED DESCRIPTION:
Background:

Juvenile idiopathic arthritis (JIA) is a heterogeneous group of diseases which encompasses all forms of arthritis of unknown etiology lasting for at least 6 weeks and with onset before the age of 16. The International League of Associations for Rheumatology (ILAR) has defined seven subtypes of JIA.

Understanding of the JIA pathogenesis over the last two decades have revolutionized therapy, reduced morbidity, and improved quality of life for those affected . Various autoantibodies have been associated with JIA, including anti-nuclear antibodies (ANA), rheumatoid factor (RF), anti-citrullinated protein autoantibodies (ACPA), and others. Although the ANA test is not used to diagnose JIA, it is of high prognostic value with respect to the risk of uveitis. ANA positivity among the JIA subtypes is the highest in patients with oligoarticular JIA (up to 70%) and is particularly more prevalent in young, female patients. The prevalence of RF in patients with JIA is very low (< 5%), and it confers a worse prognosis. In particular, RF-positive polyarticular patients are at higher risk of a more aggressive disease course and bone erosion. ACPA positive children with JIA are recommended for earlier and more aggressive therapy. Nevertheless, the diagnosis of JIA still depends mainly on clinical characteristics, imaging examination, and exclusion of other, more common causes of persistent arthritis with low serological support. Therefore, it is necessary to establish alternate methods or discover new biomarkers to further improve precise JIA diagnosis at the early stage of the disease.

Lubricin, encoded by the proteoglycan 4 (PRG4) gene, is a mucin-like molecule and includes proline, serine and threonine that provides a scaffold for glycosylation, high viscosity and low friction . It is suggested to have protective effects against synovial hyperplasia and cartilage deterioration in the joint spaces. Experimental models of osteoarthritis showed that lubricin retards cartilage degeneration, enhances cartilage repair and reduces chondrocyte apoptosis.Lubricin levels were also diminished in synovial fluid of inflammatory arthritis. Furthermore, lubricin was recently suggested to act as an antagonist for Toll like receptor (TLR 2)and (TLR 4), preventing its activation in inflammatory arthritis.Moreover, a recent study proposed a new mechanism of lubricin, including inhibition of interleukin 1β (IL-1β) and tumor necrosis factor-α (TNF-α) via CD44 binding.

Survivin is an anti-apoptotic oncoprotein, known as a tissue marker of cancer. During recent years, the role of survivin in non-malignant cells was intensively explored. Survivin has been shown essential for the differentiation, growth, and regeneration of healthy tissues. Due to its role in apoptosis and proliferation, it plays important roles in the pathogenesis of autoimmune diseases. At the preclinical phase of JIA, high levels of survivin correlate with cytokines and anticipate the formation of aggressive T helper cells (Th1) and (Th17) cells. In patients after JIA diagnosis, survivin predicts joint destructive course of the disease and resistance to anti-rheumatic treatment. Survivin has been suggested as a predictive marker of a severe course of adult RA and could be used for preclinical recognition of the disease. Survivin positive patients have poor outcomes if treated with methotrexate (MTX) monotherapy. A decrease in serum survivin concentration is associated with a better clinical response to treatment.

Compared to clinical examination and conventional radiology, musculoskeletal ultrasound (MSUS) is a more sensitive method for detecting synovitis, tenosynovitis, and erosive bone disease. In JIA, MSUS is helpful in the detection of subclinical synovitis, early diagnosis, patient classification, disease activity monitoring, determining disease remission, and guiding intra-articular injections. MSUS is a suitable imaging modality for children as it requires neither sedation nor general anesthesia and no ionizing radiation, is easily repeated, compares between joints, and allows dynamic study and multisite assessment in the same session Despite therapy advances in JIA, patients can achieve only symptoms alleviation but cannot be completely cured. Therefore, exploring the pathogenesis of the rheumatoid process is of high importance for developing precise, personalized treatments and new drug targets.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes less than 16 years at onset of disease and diagnosed with oligoarticular and polyarticular JIA, fulfilling the ILAR classification criteria of JIA, The patients will be divided according to the subtypes of JIA disease.
* Control group will include age-and-sex-matched apparently healthy children.

Exclusion Criteria:

* Patients having associated neurological or disabling diseases.
* Patients with diabetes mellitus, acute or chronic infections.
* Patients with another types of JIA other than oligoarticular and polyarticular JIA (due to different patterns and diagnostic criteria of these types of JIA)
* Patients with another causes of arthritis other than JIA

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: This study will be conducted on JIA patients recruited from the Rheumatology inpatient and outpatient clinic at Assiut University Children Hospital
Sampling Method: Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
To assess Lubricin in the serum and in the synovial fluid if available in JIA patients. | 2 months
  Lubricin will be assessed in a serum sample that will be collected from JIA patients and controls and if possible from a synovial fluid sample that will be obtained from swollen joints from patients with active disease state. The serum and synovial fluid
To assess Survivin in the serum and in the synovial fluid if available in JIA patients. | 2 months
  Survivin will be assessed in a serum sample that will be collected from JIA patients and controls and if possible from a synovial fluid sample that will be obtained from swollen joints from patients with active disease state.
  The serum and synovial fluid samples will be centrifuged and stored at - 80 °C. and the concentration of survivin and lubricin will be determined by a enzyme-linked immunoassay (ELISA test) in the serum and matched synovial fluid samples of patients with JIA and in the serum of children from the control group, by commercially available kits(rabbit anti-human survivin; R&D, no DSV00, Lille,France).
To perform MSUS on the involved joints. | 4 months
  MSUS will be done to JIA patients to detect:
  A. Synovitis: presence of joint effusion and/or synovial hypertrophy Synovitis will be graded using score from 0 to 3. 0 no synovitis
  1. minimal synovitis in joint recess up to the joint capsule.
  2. synovitis in the entire joint recess causing bulging of the joint capsule.
  3. synovitis in joint recess with bulging of the joint capsule and extension to at least one bone diaphysis. B. Blood flow: defined by defined by the presence of PD signal performed only in areas where synovitis will be detected PDUS will be graded using score from 0 to 3.
  0 no signs of vascularization.
  1. mild (single/vessel dots).
  2. moderate (confluent vessel dots in < of the synovial area).
  3. marked (confluent vessel dots in ≥ of the synovial area). The sum of grey scale (GS) and power Doppler (PD) as GSPD will be calculated. The joint with the highest GSPD will be selected as the indicator joint.

SECONDARY OUTCOMES:
To assess disease activity using Juvenile arthritis disease activity score in 27 joints (JADAS 27) in the studied JIA patients. | 3 months
  The JADAS includes the following four measures:
  * Physician's global assessment of disease activity, measured on a 0-10 visual analog scale (VAS) where 0 = no activity and 10 = maximum activity;
  * Parent global assessment of well-being, measured on a 0-10 VAS where 0 = very well and 10 = very poor
  * The erythrocyte sedimentation rate (ESR), normalized to a 0 to 10 scale according to the following formula (ESR(mm/hr)-20/10) ESR values 20 mm/hr are given 0 points ESR values 120 mm/hr are given 10 points
  * Count of joints with active disease. JADAS27 includes a selected count of the following joints: cervical spine, elbows, wrists, metacarpophalangeal joints (from first to third), proximal interphalangeal joints, hips, knees and ankles.
To identify the prevalence of functional disability in JIA children and adolescents using the childhood health assessment questionnaire (CHAQ). | 3 months
  Childhood Health Assessment Questionnaire (CHAQ) :
  Describes the child's usual activities in eight domains over the past week. It include dressing, getting up, eating, walking, hygiene, reaching overhead objects, grip and activities. Each question is scored from 0 to 3 (0 = no difficulty, 1 = some difficulty, 2 = much difficulty and 3 = unable to do). The score for each of the eight functional areas will be averaged to calculate the disability index. Patients will be classified as mildly disabeled (score >1) , moderately disabeled ) score 1-2) or severely disabeled (score <2) .

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed G Mohamed, Ass prof, Study Director — Assiut University; Manal M Ahmed, Ass prof, Study Director — Assiut University; Nagwa A Mohamed, Prof, Study Director — Assiut University

REFERENCES:
- [Background] Lipinska J, Kaszkowiak M, Malachowska B, Swidrowska-Jaros J, Smolewska E. Concentration of survivin in children with oligo- and polyarticular juvenile idiopathic arthritis (JIA): diagnostic and prognostic value-a single-center study. Arthritis Res Ther. 2021 Jan 26;23(1):40. doi: 10.1186/s13075-021-02424-y. PMID 33494811
- [Background] Mosa DM, Abdelrahman AM, El-Bahnasawy AS. Ultrasound Features across Subtypes of Juvenile Idiopathic Arthritis. Rheumato. 2022;2(1):2-14.
- [Background] Ekinci RMK, Balci S, Coban F, Bisgin A. Serum lubricin levels in patients with juvenile idiopathic arthritis. Reumatologia. 2021;59(6):373-377. doi: 10.5114/reum.2021.111696. Epub 2021 Dec 9. PMID 35079181
- [Background] Petty RE, Southwood TR, Manners P, Baum J, Glass DN, Goldenberg J, He X, Maldonado-Cocco J, Orozco-Alcala J, Prieur AM, Suarez-Almazor ME, Woo P; International League of Associations for Rheumatology. International League of Associations for Rheumatology classification of juvenile idiopathic arthritis: second revision, Edmonton, 2001. J Rheumatol. 2004 Feb;31(2):390-2. No abstract available. PMID 14760812
- [Background] Consolaro A, Giancane G, Schiappapietra B, Davi S, Calandra S, Lanni S, Ravelli A. Clinical outcome measures in juvenile idiopathic arthritis. Pediatr Rheumatol Online J. 2016 Apr 18;14(1):23. doi: 10.1186/s12969-016-0085-5. PMID 27089922
- [Background] Consolaro A, Ruperto N, Bazso A, Pistorio A, Magni-Manzoni S, Filocamo G, Malattia C, Viola S, Martini A, Ravelli A; Paediatric Rheumatology International Trials Organisation. Development and validation of a composite disease activity score for juvenile idiopathic arthritis. Arthritis Rheum. 2009 May 15;61(5):658-66. doi: 10.1002/art.24516. PMID 19405003
- [Background] Elsayed Mostafa W, Bakry Abdul-sattar A, Abo Elsaud Dawa G. Prevalence and factors of functional disability in patients with juvenile idiopathic arthritis. Zagazig University Medical Journal. 2019;25(3):456-63.
- [Background] Miotto E Silva VB, Mitraud SAV, Furtado RNV, Natour J, Len CA, Terreri MTSELRA. Patients with juvenile idiopathic arthritis in clinical remission with positive power Doppler signal in joint ultrasonography have an increased rate of clinical flare: a prospective study. Pediatr Rheumatol Online J. 2017 Nov 13;15(1):80. doi: 10.1186/s12969-017-0208-7. PMID 29132381
- [Background] Huang YH, Hu YC, Liao CH, Chiang BL, Lu CH, Li KJ, Yang YH. Utilizing ultrasound findings of a single indicator joint to assess non-systemic juvenile idiopathic arthritis. Pediatr Rheumatol Online J. 2021 Apr 29;19(1):60. doi: 10.1186/s12969-021-00550-0. PMID 33926518